CLINICAL TRIAL: NCT01852513
Title: Allergic Rhinitis Changes the Sinus Microbiome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB 12-1812
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QNASL nasal spray (Active Comparator): QNASL 320 mcg once-daily administered as two sprays in each nostril; 2 weeks of treatment
  Interventions: Drug: QNASL
- Placebo nasal spray (Placebo Comparator): Placebo nasal spray once-daily administered as two sprays in each nostril; 2 weeks of treatment
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: QNASL
  Arms: QNASL nasal spray
Drug: Placebo nasal spray
  Arms: Placebo nasal spray

SUMMARY:
The investigators hypothesize that treatment with QNASL will reduce nasal mucosal inflammation induced by the allergy season and prevent the changes in the microbiome caused by the allergy season.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 55 years of age.
2. Two year history of seasonal allergic rhinitis.
3. Positive skin test to grass and/or tree antigen.

Exclusion Criteria:

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Subjects treated with systemic steroids during the previous 30 days.
4. Subjects treated with topical (inhaled, intranasal or intraocular) steroids, Nasalcrom or Opticrom during the previous 30 days.
5. Subjects treated with oral antihistamine/decongestants during the previous seven days.
6. Subjects treated with topical (intranasal or intraocular) antihistamine/decongestants during the previous 3 days.
7. Subjects treated with immunotherapy and are escalating their dose.
8. Subjects on chronic anti-asthma medications.
9. Subjects with polyps in the nose or a significantly displaced septum.
10. Upper respiratory infection within 14 days prior to study start.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Pinto, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- QNASL Nasal Spray: QNASL 320 mcg once-daily administered as two sprays in each nostril; 2 weeks of treatment
  QNASL
- Placebo Nasal Spray: Placebo nasal spray once-daily administered as two sprays in each nostril; 2 weeks of treatment
  Placebo nasal spray
Period: Overall Study
Arm/Group | QNASL Nasal Spray | Placebo Nasal Spray
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QNASL Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Total Nasal Symptom Score (TNSS)
Description: The Total Nasal Symptom Score (TNSS) is the sum of scores for each of nasal congestion, sneezing, nasal itching, and rhinorrhea using a four point scale (0-3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. TNSS is calculated by adding the score for each of the symptoms to a total out of 12. TNSS was assessed daily and summed over 14 days; thus, the total score ranges from 0 to 168, with higher scores indicating a worse outcome.
Time Frame: Two weeks following initiation of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QNASL Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 20 | 19
score on a scale | 67.1 (43.2) | 78.0 (34.3)
Statistical Analysis 1: Comparison: QNASL Nasal Spray vs Placebo Nasal Spray; Test type: Superiority; p = 0.391, t-test, 2 sided

2. Primary Outcome: Change in RQLQ Score From Baseline to Two Weeks
Description: The Rhinoconjunctivitis Quality Of Life Questionnaire (RQLQ) is a self-administered disease-specific health-related quality of life instrument that measures the functional impairments that are most troublesome to adult patients as a result of their seasonal or perennial rhinoconjunctivitis of either allergic or non-allergic origin. There are 28 items each asking about symptoms during the previous week. Seven domains of activity limitation are included: activities (3 "patient-specific") limitation, sleep problems (3 items), nose symptoms (4 items), eye symptoms (4 items), non-nose/eye symptoms (7 items), practical problems (3 items) and emotional function (4 items)). Each item is reported using a 7-point scale (0 = not impaired at all, 6 = severely impaired), and a total score is calculated by averaging over all items (range 0-7). Higher scores reflect lower quality of life.
Time Frame: Two weeks following initiation of treatment
Population: Those analyzed included all participants with data for this measure at baseline and two weeks.
Measure: Mean (Standard Deviation); unit: Change in scale score
Arm/Group | QNASL Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 20 | 18
Change in scale score | 1.2 (1.1) | 1.3 (1.3)
Statistical Analysis 1: Comparison: QNASL Nasal Spray vs Placebo Nasal Spray; Test type: Superiority; p = 0.789, t-test, 2 sided

3. Primary Outcome: Change in Percent Eosinophils From Baseline to Two Weeks
Description: The percentage of nasal eosinophils recovered from nasal lavage was assessed at baseline and after two weeks of treatment.
Time Frame: Two weeks following initiation of treatment
Population: Those analyzed included all participants with data for this measure at baseline and two weeks.
Measure: Mean (Standard Deviation); unit: Change in percentage of eosinophils
Arm/Group | QNASL Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 8 | 8
Change in percentage of eosinophils | 1.5 (3.5) | 2.1 (4.8)
Statistical Analysis 1: Comparison: QNASL Nasal Spray vs Placebo Nasal Spray; Test type: Superiority; p = 0.778, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Two weeks following initiation of treatment
Arm/Group | QNASL Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No